CLINICAL TRIAL: NCT03625089
Title: The Impact of Nurse-led Programme With and Without Carotid Ultrasound on Addressing Cardiovascular Risk in Patients With Arthritis: a Prospective, Multicentre, Randomised, Controlled Trial
Brief Title: Impact of Nurse-led Programme With Carotid Ultrasound on Addressing Cardiovascular Risk in Patients With Arthritis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited funding support
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IA_2017
Record Dates: First submitted 2018-07-04; First posted 2018-08-10 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Arthritis, Rheumatoid; Arthritis, Psoriatic
Keywords: Carotid Atherosclerosis; Arterial Stiffness; Cardiovascular Risk
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Carotid Artery Diseases | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - FRS arm (Active Comparator): Both group will participate in the nurse-led programme on CV risk screening and carotid ultrasound for carotid plaque assessment. Subjects in group 1 will initiate Atorvastatin treatment (20mg daily per oral) if their Framingham Risk Score >10%
  Interventions: Drug: Atorvastatin
- Group 2 USG arm (Experimental): Subjects in group 2 will initiate Atorvastatin treatment (20mg daily per oral) if they had carotid plaque upon carotid ultrasound findings..
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Group 1 patients will be prescribed statin when FRS > 10%; while group patients will be prescribed statin upon presence of carotid plaque as reported from carotid ultrasound. The decision will solely be made base on the randomized group by either FRS>10% or presence of carotid plaque.
  Atorvastatin 20 mg is recommended as the preferred initial high intensity statin to use because it is clinically and cost effective for the primary prevention of CVD according to the national institute for Health and Care Excellence (NICE) guideline from the United Kingdom.
  Other Names: Lipitor

SUMMARY:
Elevated CVD risk is a significant public health problem that contributes greatly to the increased morbidity and shortened lifespan of individuals with RA and PsA. Over the past decades, there has been great progress into the understanding of the severity of CVD risk in these patients but these risk factors are not well managed. The development of the high-risk strategy is therefore necessary, with more intensive therapy reserved for patients identified as high-risk, e.g. because they have high-risk FRS. However, these risk scores under-estimated CV risk in patients with RA and PsA. An intermediate approach is to use quantification of preclinical vascular disease to further identify high-risk patients. Results from this study will provide clinical implications in terms of detecting and managing cardiovascular morbidity in patients with RA and PsA.

DETAILED DESCRIPTION:
Objectives This study investigates the impact of a nurse-led programme on cardiovascular (CV) risk screening with and without carotid ultrasound for carotid plaque on CV risk factor control in asymptomatic rheumatoid arthritis (RA) and psoriatic arthritis (PsA) patients.

Hypothesis The investigators hypothesize that CV risk stratification and management in RA and PsA may be improved by incorporation of carotid ultrasound to assess for carotid plaque.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RA fulfilled the 2010 ACR/EULAR classification criteria or PsA fulfilled the Classification of Psoriatic Arthritis (CASPAR) criteria
* aged between 18 and 75 will be recruited.

Exclusion Criteria:

* had a history of overt CVD (ie, symptomatic coronary artery disease [CAD] or ischemic stroke or transient ischemic attack or peripheral vascular disease)
* had significant co-morbidities including severe renal impairment or severe deranged liver function
* female of childbearing potential who are unwilling to use adequate contraception, pregnant or breastfeeding women
* patients who are already taking lipid lowering therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
change in Framingham risk score | 12 months
  The Framingham Risk Score is a gender-specific algorithm used to estimate the 10-year cardiovascular risk of an individual. Individuals with low risk have 10% or less CHD risk at 10 years, with intermediate risk 10-20%, and with high risk 20% or more. Change in Framingham risk score between subject in two group will be evaluated. A positive change in score indicates increased CV risk, vice versa.

SECONDARY OUTCOMES:
Change in pulse wave velocity (PWV) in subjects | 12 months
  Change in arterial stiffness in terms of PWV (cm/s) in subjects between subject in two group, as a parameter to capture change in CV risk upon intervention
Change in augmentation index (AIX) in subjects | 12 months
  Change in arterial stiffness in terms of AIX (%)in subjects between subject in two group, as a parameter to capture change in CV risk upon intervention
Change in individual modifiable risk factors levels | 12 months
  Target for individual modifiable risk factor will be set (For subject with diabetes, target is Hba1c<7.0%; for dyslipidaemia subject, target is LDL<2.6 mmol/l; for obese subject, target is drop in BMI for 1 unit; for smoker, target is smoking cessation; for all subject, physical activity level target is at least once per week with not less than 30 min activity) Change total number of modifiable risk factor achieved target will be computed.
The number of measures taken against comorbidities | 12 months
  The number of measures taken against commodities (including home blood pressure monitoring, attending dietitian education class, compliance to drug etc) after implementation of nurse led clinic
Proportions of patients achieving remission | 12 months
  Proportions of patients achieving remission between two group to evaluate outcome upon treat-to-target protocol
Changes in intima-media thickness (IMT) | 12 months
  Changes in IMT (mm) in subjects between 2 groups after intervention by using high-resolution ultrasound
Proportion of plaque progression | 12 months
  Proportion of plaque progression in subjects between 2 groups after intervention by using high-resolution ultrasound.
  Plaque progression defined as increase in area harboring plaque or increased number of plaque

CONTACTS AND LOCATIONS:
Overall Officials: Lai Shan Tam, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine and Therapeutics, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT03625089/Prot_000.pdf